CLINICAL TRIAL: NCT06660095
Title: "Investigation of the Clinical Predictive Value of p50 Value in Liver Transplant Surgeries"
Brief Title: Intraoperative "p50" Measurement in Liver Transplant Surgeries
Acronym: p50
Status: Enrolling by invitation | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yusuf Ziya ÇOLAK, Assoc. Prof. Muharrem Ucar, MD., Inonu University
Other Study IDs: Inonu p50
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplant; Complications
Keywords: Liver transplant; anesthesia; Blood gas analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant recipients: T0: After the anesthesia induction, before the surgery T1: Intraoperative p50 value from the blood gas sample taken during the dissection stage T2: Intraoperative p50 value from the blood gas sample taken during the anhepatic stage T3: Intraoperative p50 value from the blood gas sample taken during the neohepatic stage T4: After the hepatic artery reperfusion T5: At the end of the surgery

SUMMARY:
The aim of this study is to compare the p50 value in routine blood gas measurements taken during liver transplant surgery follow-up with other follow-up parameters and clinical findings on the monitors, and to investigate whether there is a predictive parameter that can predict the rapidly changing clinical findings of the patients.

DETAILED DESCRIPTION:
Blood gas monitoring is the most commonly method used by anesthetists during liver transplant surgeries. We evaluated the blood gas p50 value according to the stages in these heart transplant operations. We tried to find out how the blood gas p50 value would guide the patient's clinical findings in the dissection phase, anhepatic phase and neohepatic phase. For this purpose, we compared arterial and venous blood gas p50 values with the patient's vital signs at certain stages in liver transplant surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients who will undergo Elective Liver Transplant surgery at İnönü University Faculty of Medicine Liver Transplant Institute, ASA (American Society of Anesthesiology) score III-IV, patients between the ages of 18-65

Exclusion Criteria:

* Patients with fulminant liver failure,
* hepatic encephalopathy,
* hepatorenal,
* hepatopulmonary syndrome,
* uncontrolled diabetes mellitus,
* cardiovascular, pulmonary disease,
* sepsis
* and patients who refuse consent in the informed consent form will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant recipients who will undergo Elective Liver Transplant surgery at İnönü University Faculty of Medicine Liver Transplant Institute, ASA (American Society of Anesthesiology) score III-IV, patients between the ages of 18-65
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-12-21 (Estimated); Study Completion 2025-01-21 (Estimated)

PRIMARY OUTCOMES:
p50 changes during liver transplant surgery | T0: at the end of the dissection before clamps T1: 5 min. before reperfusion (anhepatic) T2: 30 min. after reperfusion of the liver graft (neohepatic) T3: after hepatic artery reperfusion T4: End of the operation
  P50 is the partial pressure of oxygen required to achieve 50% haemoglobin saturation. The normal p50 value is 24-28 mmHg. The oxygen-hemoglobin dissociation curve represents the affinity of hemoglobin for oxygen. The p50 value represents a mid-point in this curve, and gives us information regarding that affinity. Determining the clinical value, if any, of the changes in p50 values taken at different stages of liver transplantation surgery may be useful in the follow-up of these patients in the future and may help in making intraoperative decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Muharrem UCAR, assoc.Prof., Study Director — Inonu University
Locations (1):
- İnönü Üniversitesi Merkez Kampüsü (Elazığ Yolu 15.km) Battalgazi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim Y, Jung JH, Kim GE, Park M, Lee M, Kim SY, Kim MJ, Kim YH, Kim KW, Sohn MH. P50 implies adverse clinical outcomes in pediatric acute respiratory distress syndrome by reflecting extrapulmonary organ dysfunction. Sci Rep. 2022 Aug 11;12(1):13666. doi: 10.1038/s41598-022-18038-6. PMID 35953629
- [Result] Hall TH, Dhir A. Anesthesia for liver transplantation. Semin Cardiothorac Vasc Anesth. 2013 Sep;17(3):180-94. doi: 10.1177/1089253213481115. Epub 2013 Mar 12. PMID 23482506